CLINICAL TRIAL: NCT05114993
Title: End-tidal Carbon Dioxide Measurements in Adults and Children Wearing Surgical Masks
Brief Title: The Effect of Wearing Masks on End-tidal Carbon Dioxide and Pulse Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Brooks (Other)
Collaborators: Missouri State University (Other)
Responsible Party: Sponsor-Investigator, Patrick Brooks, Assistant Professor, Missouri State University
Organization: Missouri State University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CT-2021-01
Record Dates: First submitted 2021-10-18; First posted 2021-11-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Carbon Dioxide
Keywords: surgical masks; end tidal CO2; pulse oximetry

STUDY DESIGN:
Intervention Model Description: Participants will be observed and monitored for 5 minutes without any intervention. After 5 minutes of observation and monitoring, participants will don a disposable surgical mask. Participants will then be observed and monitored for 15 minutes while under the intervention of "mask-wearing". Only one type of mask will be used for all participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of donning a disposable surgical mask (Experimental): Participants will be observed and monitored without wearing a mask for a 5-minute control period. Measurements will include End Tidal CO2, Inspired CO2, Pulse Oximetry, Respiratory Rate, and Heart Rate each minute without a mask x 5 minutes.
  After 5 minutes, all study subjects will don the same model of disposable surgical mask. The same measurements will be taken, including End Tidal CO2, Inspired CO2, Pulse Oximetry, Respiratory Rate, and Heart Rate each minute with a mask x 15 minutes.
  Interventions: Device: wearing a disposable surgical mask

INTERVENTIONS:
Device: wearing a disposable surgical mask — Physiologic vital signs will be monitored every minute for 5 minutes without a mask, followed by every minute for 15 minutes with a surgical mask.

SUMMARY:
An Interventional Study is planned with the primary purpose of screening for changes in end-tidal carbon dioxide (ETCO2), inspired carbon dioxide (ICO2), and other vital signs that may develop after donning a disposable surgical mask.

Measurements will be taken and recorded during a 5-minute control period without a mask, recording non-invasive ETCO2 and ICO2 levels by way of a nasal cannula (NC), oxygen saturation (SpO2), breaths per minute (RR), and heart rate (HR) via anesthesia equipment. This will be followed by a 15-minute intervention of wearing a disposable surgical mask and repeating measurements of ETCO2, ICO2, SpO2, RR, and HR, recorded each minute.

Data will be collected from adults and children as young as 2 years of age. Age groups will include children aged 2-14 and adults aged 18 to 80, as described in the details of the research protocol. Parents and their children are invited to participate together.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Aged 2 - 14 years (inclusive) or 18 - 80 years (inclusive)

Exclusion Criteria:

* Significant cardiopulmonary diseases
* Intolerance to wearing nasal canula
* Intolerance to wearing a surgical mask

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Potential Change in End Tidal CO2 level | End tidal CO2 levels after 5 minutes without a mask will be compared to End Tidal CO2 levels after 15 minutes wearing a disposable surgical mask
  measurement of End Tidal CO2 by way of nasal cannula

SECONDARY OUTCOMES:
Potential change in Inspired CO2 level | Inspired CO2 levels after 5 minutes without a mask will be compared to Inspired CO2 levels after 15 minutes wearing a disposable surgical mask
  measurement of inspired CO2 by way of nasal cannula
Potential change in oxygen saturation | Oxygen saturation levels after 5 minutes without a mask will be compared to oxygen saturation levels after 15 minutes wearing a disposable surgical mask
  measurement of oxygen saturation by way of noninvasive pulse oximetry
Potential change in respiratory rate measured in breaths per minute | Respiratory rate after 5 minutes without a mask will be compared to respiratory rate after 15 minutes wearing a disposable surgical mask
  measurement of breaths per minute
Potential change in Heart Rate | Heart rate after 5 minutes without a mask will be compared to heart rate after 15 minutes wearing a disposable surgical mask
  measurement of heart rate in beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri State University, Springfield, Missouri, United States

REFERENCES:
- [Derived] Brooks JP, Layman J, Willis J. Physiologic effects of surgical masking in children versus adults. PeerJ. 2023 Jun 16;11:e15474. doi: 10.7717/peerj.15474. eCollection 2023. PMID 37342359